CLINICAL TRIAL: NCT06678958
Title: Intermediate Term Outcomes of Trabecular Metal Augments Used in the Flying Buttress Position in the Management of Acetabular Defects
Brief Title: Outcomes of Trabecular Metal Augments Used in the Flying Buttress Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tony Maher, Lecturer of orthopedic surgery, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trabecular metal augments
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Acetabular Abnormality
Keywords: Acetabular augments; Flying buttress; Revision total hip replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult patients with acetabular defects requiring reconstruction (Experimental): The acetabular defect was reconstructed by tarbecular metal augments in the flying buttress position
  Interventions: Procedure: Reconstruction of acetabular defect by trabecular metal augment

INTERVENTIONS:
Procedure: Reconstruction of acetabular defect by trabecular metal augment — The augments were used in the flying buttress position

SUMMARY:
This study hypothesize that trabecular metal augments used in the flying buttress position is a valid option with good results in the management of uncontained acetabular defects.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* 18 years or older
* acetabular defect paprosky 2b or 3a segemntal defect reconstructed with trabecualr metal augment in the flying buttress position.

Exclusion Criteria:

* patients presented with active infection
* pathological defects
* pelvic discontinuity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Functionl hip status | 8 years
  Functional outcome was assessed by oxford hip score the worst score is 12 and the best score is 60
Survivorship of the construct | 8years
  The rate of construct survivorship using the kaplan meier survival analysis